CLINICAL TRIAL: NCT01871623
Title: Stability of One-Piece Le Fort I Osteotomy Versus Segmental Le Fort I Osteotomy: A Prospective Study
Brief Title: One-Piece Le Fort I Osteotomy Versus Segmental Le Fort I Osteotomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 101-4416A3
Record Dates: First submitted 2013-05-23; First posted 2013-06-07 (Estimated); Last update posted 2013-06-07 (Estimated); Status verified 2013-03

CONDITIONS: Cleft Lip and Palate; Le Fort
Keywords: Cleft lip and palate; Cone-Beam Computed Tomography; Le Fort I Osteotomy; Segmental Osteotomy; Stability
MeSH Terms: conditions — Cleft Lip

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Segmental Le Fort I Osteotomy (Experimental): For some cases that bone filling over cleft site is not good enough for tooth movement, it is possible that we put them into this group which means by using Segmental Le Fort I Osteotomy to approximate two dental alveolar segments.
  Interventions: Procedure: Segmental Le Fort I osteotomy
- One-piece Le Fort I Osteotomy (Active Comparator): For patients having ideal bone graft result over cleft site, traditional One-piece Le Fort I Osteotomy will be performed.
  Interventions: Procedure: One-piece Le Fort I Osteotomy

INTERVENTIONS:
Procedure: Segmental Le Fort I osteotomy — comparison the stability of segmental Le Fort I osteotomy with conventional approach of one-piece Le Fort I osteotomy
  Other Names: Segmental maxillary osteotomy; Maxillary Segmental osteotomy
  Arms: Segmental Le Fort I Osteotomy
Procedure: One-piece Le Fort I Osteotomy — conventional approach
  Other Names: Le Fort I Osteotomy; Le Fort 1 Osteotomy
  Arms: One-piece Le Fort I Osteotomy

SUMMARY:
Le Fort I osteotomy is often used in orthognathic surgery for patients to solve midface retrusion. It is known that post-surgical stability of Le Fort I osteotomy can be influenced by single jaw or bimaxillary procedures, fixation techniques or interpositional grafting. In patients with cleft lip and palate, the postoperative instability of Le Fort I osteotomy can be even worse due to scar tissue resulted from palate surgery. Segmental LeFort I osteotomy is another useful surgical modifications that can be easily done through the alveolar cleft. It is performed to allow the correction of differences in the occlusal planes, correction of transverse discrepancy or to facilitate an optimal occlusion. The most important benefits is that the alveolar cleft in patients who have not had alveolar bone graft surgery or failed to have successful result can be narrow down or even closed by approximation of two separating alveolar segments. However, there are limited previous studies comparing the stability of segmental versus one-piece Le Fort I osteotomy especially in patients with cleft. It is our aim to investigate whether one-piece Le Fort I osteotomy or segmental Le Fort I osteotomy can provide a better stability after surgery.

DETAILED DESCRIPTION:
Measurements Skeletal movement

1. Skeletal Surgical movement from T2 to T1

   * positional change of landmarks in vertical from constructed Frankfurt plane
   * positional change of landmarks in horizontal plane in relative to constructed coronal plane through Sella point
2. Post-Surgical skeletal movement (Stability) from T3 to T2

   * positional change of landmarks in vertical from constructed Frankfurt plane
   * positional change of landmarks in horizontal plane in relative to constructed coronal plane through Sella point
3. Skeletal angular measurement change on mid-sagittal plane from (T2 to T1) and (T3 to T2)
4. Dental change measured from digital maxillary cast in transverse direction from (T2 to T1) and (T3 to T2)
5. Facial Height / Facial Proportion changes from (T2 to T1) and (T3 to T2)
6. Alveolar cleft width changes from (T2 to T1) and (T3 to T2)

ELIGIBILITY:
Inclusion Criteria:

1. Cleft lip/palate patients
2. Non growing Taiwanese adults, at least 18 years old for men and 16 years old for women
3. Patients with midface retrusion and malocclusion that will need Le Fort I osteotomy
4. Rigid fixation with bone plates
5. Patients who signs the informed consent form

Exclusion Criteria:

1. Association with craniofacial anomalies
2. Patient without complete 3D imaging records including CBCT scans and digital dental models

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-04; Primary Completion 2016-03 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
stability and relapse rate of surgical movement | 6 months after surgery & 1-2 years till the completion of the treatment
  to compare the stability and relapse rate in vertical, horizontal and transverse among two kinds of different surgical techniuques

SECONDARY OUTCOMES:
Presence of pathological change of cleft-adjacent teeth | immediate after surgery, 6 months after surgery & 2 years till the completion of the treatment
  record any periodontal breakdown or periapical radiolucency of cleft-adjacent teeth

CONTACTS AND LOCATIONS:
Overall Officials: Yu Fang Liao, Ph.D., Study Director — Chang Gung Craniofacial Center , Chang Gung Memorial Hospial , Taoyuan , Taiwa
Locations (1):
- Chang Gung Craniofacial Center, Taipei / Taoyuan, Taiwan